CLINICAL TRIAL: NCT06991244
Title: The Effectiveness of EMDR 2.0 Group Intervention on Post-Traumatic Stress, Depression, and Anxiety Symptoms in Earthquake Survivors
Brief Title: EMDR 2.0 Group Therapy for PTSD, Depression, and Anxiety in Earthquake Survivors
Acronym: EQ-EMDR20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Çiğdem Kınık, Principal Investigator, PhD Researcher in Applied Psychology, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KINIK EMDR 2.0 EQ
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Post-Traumatic Stress Disorder (PTSD); Depression; Anxiety
Keywords: PTSD; Depression; Anxiety; Disaster; Earthquake; EMDR 2.0; Group Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR 2.0 Group (Experimental): Participants in this group received a face-to-face EMDR 2.0 group intervention delivered over three sessions in a container city setting in Malatya, Türkiye, following the 2023 earthquake.
  Interventions: Behavioral: EMDR 2.0 Group Protocol
- Control Group (No Intervention): Participants in this group did not receive any psychological intervention during the study period but completed the same assessments as the intervention group.

INTERVENTIONS:
Behavioral: EMDR 2.0 Group Protocol — A short-term trauma-focused group protocol adapted from EMDR 2.0, delivered in three sessions over one week, targeting PTSD, depression, and anxiety symptoms among earthquake survivors. The first session lasted 90 minutes, followed by two 60-minute sessions. The intervention was administered face-to-face in a container city in Malatya, Türkiye. All sessions were conducted by a certified EMDR therapist who had completed advanced EMDR 2.0 training.
  Arms: EMDR 2.0 Group

SUMMARY:
The objective of this clinical study was to examine whether a brief EMDR 2.0 group intervention could reduce symptoms of post-traumatic stress disorder (PTSD), depression, and anxiety in adult survivors of the 2023 Türkiye earthquake. The study was conducted face-to-face in a container city in Malatya, one of the regions most severely affected by the disaster. EMDR 2.0 is an enhanced version of standard EMDR therapy that uses working memory taxation techniques to accelerate emotional processing.

The primary research questions included whether EMDR 2.0 group therapy reduces PTSD symptoms in earthquake survivors, and whether it helps decrease symptoms of depression and anxiety.

Participants attended three EMDR 2.0 group sessions in person over the course of one week and completed psychological assessments before the intervention, one week after, and one month after. Verbal disclosure of traumatic memories was not required during the sessions. Researchers used self-report questionnaires to evaluate changes in trauma-related distress, depression, and anxiety. This study contributes to the development of fast, accessible, and field-based psychological support strategies for communities affected by disasters.

DETAILED DESCRIPTION:
Following the 2023 Türkiye earthquakes, widespread displacement, loss, and psychological trauma created an urgent need for effective and accessible mental health interventions. This clinical study was developed to address that need by offering a rapid, structured group therapy protocol-EMDR 2.0-to adult survivors residing in a temporary container city in Malatya, a region significantly impacted by the disaster.

EMDR 2.0 is a modified version of traditional Eye Movement Desensitization and Reprocessing therapy. It intensifies working memory taxation through structured, dual-attention tasks and allows for the safe and efficient processing of traumatic memories without requiring verbal disclosure.

The intervention was delivered in the same container units used as temporary housing by survivors, thereby transforming these living spaces into short-term therapeutic settings. Over the course of one week, three group sessions were administered in person. While participants were gathered in a group format, each individual engaged in processing their own traumatic imagery using the EMDR 2.0 protocol.

This approach provided containment and emotional safety within a physically and psychologically shared post-disaster context. Verbal expression of trauma was not required, which minimized the risk of retraumatization and enhanced the accessibility of the intervention for individuals hesitant to disclose.

The study was designed not only to evaluate the effectiveness of EMDR 2.0 in reducing symptoms of PTSD, depression, and anxiety but also to assess the feasibility of implementing this method under real-world post-disaster conditions with limited resources. The findings contribute to the growing body of knowledge on scalable trauma interventions suitable for use in field-based, high-need humanitarian settings.

This work underscores the potential of brief, structured group interventions to facilitate emotional recovery when survivors are supported in environments that respect both their privacy and collective experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Being a survivor of the 2023 Türkiye earthquakes
* Currently residing in a temporary container settlement in Malatya
* Ability to attend all three face-to-face intervention sessions
* Ability to provide informed consent
* Sufficient cognitive and emotional capacity to complete self-report questionnaires
* Basic literacy (reading and writing) in Turkish to understand and complete self-report scales
* Willingness to voluntarily participate in the study

Exclusion Criteria:

* Having a current diagnosis of a psychotic disorder (e.g., schizophrenia, bipolar disorder with psychotic features)
* History of severe head trauma or neurological condition affecting cognitive capacity
* Active suicidal ideation or risk requiring emergency psychiatric care
* Ongoing substance dependence
* Receiving concurrent trauma-focused psychotherapy during the study period
* Significant hearing, vision, or language impairment interfering with participation
* Inability to attend scheduled sessions or complete follow-up assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity | Assessed at three time points - before the intervention (Day 0), one week after the completion of the third session (approximately Day 7), and one month after the completion (approximately Day 30)
  The primary outcome is the change in PTSD symptoms as measured by the PCL-5, a 20-item self-report questionnaire that assesses PTSD symptoms based on DSM-5 criteria. The scale includes four subscales: intrusion, avoidance, negative alterations in cognition and mood, and alterations in arousal and reactivity. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Depression symptom severity (DASS-21 Depression subscale) | Assessed at three time points: before the intervention (Day 0), one week after completion of the third session (approximately Day 7), and one month after completion (approximately Day 30)
  The DASS-21 Depression subscale evaluates core symptoms such as dysphoria, hopelessness, and devaluation of life. Higher scores indicate more severe depressive symptoms.
Anxiety symptom severity (DASS-21 Anxiety subscale) | Assessed at three time points: before the intervention (Day 0), one week after completion of the third session (approximately Day 7), and one month after completion (approximately Day 30)
  The DASS-21 Anxiety subscale measures autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect.
Stress symptom severity (DASS-21 Stress subscale) | Assessed at three time points: before the intervention (Day 0), one week after completion of the third session (approximately Day 7), and one month after completion (approximately Day 30).
  The DASS-21 Stress subscale evaluates persistent tension, irritability, and difficulty relaxing. Higher scores indicate elevated stress-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alisan B Yasar, MD AssocProf, Study Chair — Istanbul Gelisim University
Locations (1):
- Malatya Teknokent Container Settlement, Battalgazi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study was conducted as part of a doctoral thesis project. Data sharing was not specified in the ethics committee approval. The sample is small and consists of individuals affected by a major natural disaster, living in a container settlement, making the data highly sensitive. Given the nature of the trauma-focused intervention and the emphasis on confidentiality, informed consent for IPD sharing was not obtained. Therefore, individual participant data will not be shared.